CLINICAL TRIAL: NCT05795491
Title: Effect of Blue Light Emitting Diode Therapy on Recurrent Vulvovaginal Candidiasis
Brief Title: Blue Light Emitting Diode Therapy on Vulvovaginal Candidiasis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Radwa Mohamed Reda Shalaby, Physiotherapist, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 012/004261
Record Dates: First submitted 2023-03-21; First posted 2023-04-03 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-05

CONDITIONS: Recurrent Vulvovaginal Candidiasis
MeSH Terms: conditions — Candidiasis, Vulvovaginal | interventions — Fluconazole

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Group A (Placebo Comparator): This group includes 30 patients will receive routine medical treatment with antifungal, azole (vaginal route).
  100 ml ( one Suppository ) at bedtime for three nights in a row
  Interventions: Drug: Azole Antifungal
- Group B (Experimental): This group includes 30 patients. The vulva and vagina will be exposed to 401 ± 5 nm ultraviolet A/ blue LED irradiation in a single session, divided into two applications.
  Interventions: Device: Blue Light Emitting Diode Therapy

INTERVENTIONS:
Device: Blue Light Emitting Diode Therapy — Light-emitting diode (LEDs) as a preferred light source for phototherapy is a semiconductor device that, through the process of electroluminescence, generates light emitted at different wavelengths, causing a differentiation in color and effects.
  Other Names: Blue LED
  Arms: Group B
Drug: Azole Antifungal — Azole antifungals are a group of medicines that contain an azole ring and inhibit the growth of a wide range of fungi
  Other Names: fluconazole
  Arms: Group A

SUMMARY:
With the knowledge that VVC is an infectious disease of the genitourinary tract that is common in women of reproductive age, and because of the shortage of non-drug therapies for this condition, this study will aim to evaluate the effect of ultraviolet A/blue LED with a wavelength of 401 ± 5 nm in patients with a clinical manifestation of candidiasis and its ability to prevent recurrence.

DETAILED DESCRIPTION:
Vulvovaginal candidiasis (VVC) is an infection of the vulva and vagina caused by the abnormal growth of several Candida species. This pathology is one of the most common diagnoses in gynecological practice and the second most common genital infection. Studies have shown that 15 to 25% of adult women present with fungal colonization despite being asymptomatic and that 75% of them will develop the disease at some point in their lives.

The treatment of VVC involves the use of antifungal agents, either orally or topically, which resolves 80 to 90% of the cases. However, the use of these agents can lead to the development of adverse reactions such as dysuria, pruritus, and gastrointestinal disorders.

Accordingly, a hypothesis arises that the blue/violet light- emitting diode (LED) may be an alternative treatment for women with VVC because of its antimicrobial effect that has been proven by several studies. Moreover, it is considered a safe, non-invasive, painless, and non-toxic technique for use in several types of tissue.

ELIGIBILITY:
Inclusion Criteria:

subject selection will be according to the following criteria:

1. Age will range between 18- 50 years.
2. All patients will be confirmed by culture and examination of fresh vaginal samples, to have VVC.
3. All patients who will be enrolled to the study will have their informed consent.

Exclusion Criteria:

The participants will be excluded if they meet one of the following criteria:

1. Individuals on any other antifungal drugs.
2. Individuals with cardiopulmonary conditions.
3. Individuals undergoing another radiation therapy.
4. Sensory impairment

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Vaginal swab culture . | 2 months
  It will be taken before and after the treatment and after one month for assessment of recurrence, by using a potassium hydroxide (KOH) test and fresh cytology with saline solution will be used to analyze the composition of the vaginal discharge under optical microscope

SECONDARY OUTCOMES:
Litmus Paper | 2 months
  •Litmus paper for measuring vaginal PH before and after treatment and after one month of recurrence. A vaginal pH test measures the acidity of the vagina on a scale of 1-14, by holding a piece of pH paper against the wall of your vagina for a few seconds, then compare the color of the pH paper to the color on the chart provided with the test kit. The number on the chart for the color that best matches the color on the pH paper is the vaginal pH number.

CONTACTS AND LOCATIONS:
Overall Officials: Soheir El-kosery, PHD, Principal Investigator — Professor of physical Therapy, Faculty of Physical therapy, Cairo University
Locations (1):
- Faculty of physical therapy, Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
All Data including assessment measures, treatment and results